CLINICAL TRIAL: NCT02225717
Title: Markers of Fetal Membranes Remodelling in Cervicovaginal Fluid and Delivery
Brief Title: Identification of Spontaneous Delivery Markers
Acronym: TrophY2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: P140502
Record Dates: First submitted 2014-08-07; First posted 2014-08-26 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Preterm Labor (24 GA - 32 GA)
Keywords: Preterm labor; cervicovaginal secretions; markers of fetal membranes remodelling; Multiplex test
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non pregnant women (Experimental): Healthy pregnancy : women 15-16 weeks of gestation, at 35-36 weeks of gestation, and >37 weeks of gestation and planed cesarean prior labor
  Interventions: Procedure: Cervicovaginal swab
- Preterm Labor (Experimental): Pregnant women admitted for preterm labor
  Interventions: Procedure: Cervicovaginal swab
- Healthy pregnancy (Experimental): Healthy pregnancy : women 15-16 weeks of gestation, at 35-36 weeks of gestation, and >37 weeks of gestation and planed cesarean prior labor
  Interventions: Procedure: Cervicovaginal swab

INTERVENTIONS:
Procedure: Cervicovaginal swab — Sample of cervicovaginal secretions made by the surgical team using a sterile swab introduced directly into the posterior fornix of vagina for one minute during the insertion of the urinary catheter

SUMMARY:
The investigators project aims to identify, in pregnant women, discriminating molecules to allow an early detection of women who will spontaneously deliver prematurely, suitable in routine clinical practice.

Human parturition is tightly correlated with hormonal changes at the maternal-fetal interface during pregnancy, that may control cell interactions and fetal membranes (the water bag) remodelling. Precocious remodelling may lead to a premature onset of labor, associated or not with premature rupture of membrane whether the cause is infectious or not.

In this regard, remodelled fetal membranes overlying the cervix may discharge signals that could be detectable in cervico-vaginal fluids and serve as biomarkers of the imminence of delivery. Such information on delivery timing may be of great importance for an adequate prediction that would change drastically the management of threatening preterm delivery.

DETAILED DESCRIPTION:
Prematurity is a major Public Health concern in developed countries, since it is the first cause of perinatal morbi-mortality and of cerebral palsy in early childhood. Premature birth rate has risen by 36 percent over the last 25 years to reach 7.2% in 2010 in France. Antenatal corticosteroids administration before 34 weeks and in utero transfer in high-qualified maternity wards are ones of the rare antenatal therapies recommended to improve neonatal complications of preterm delivery. Early identification of women with high risk of preterm birth should be helpful to implement those prophylactic measures. Moreover discriminating true preterm labor (PTL) vs. symptoms of PTL in women, who will finally deliver at term, would reduce unnecessary hospitalizations and prescriptions.

During human gestation, fetal membranes (the "water bag") encompass the amnion, facing the amniotic cavity, and the chorion, lining the maternal decidua and comprising trophoblast cells. Membranes usually remain intact until their spontaneous rupture, close to the first stage of labor at term. Often seen as a simple inert shell, with a role of "airbag" for the developing fetus, the membranes provide yet a large surface of interaction between maternal and fetal tissues and function as a transient endocrine organ with immune properties.

Specific remodelling of the membranes is observed at term prior to delivery. During this remodelling, drastic changes in extracellular matrix occur, with the secretion of specific molecules. The investigators hypothesize that premature fetal membranes remodelling occurs weeks prior to actual birth and may be able to be detected in women at risk for preterm birth, i.e. presenting signs of PTL. This study investigates if the detection of fetal membranes remodelling in cervico-vaginal fluids can accurately identify those women at greatest risk for preterm birth. A prospective cohort of pregnant women will before 32 weeks of gestation with symptoms of preterm labor be enrolled. As negative controls, healthy pregnant women at 12-15 or 35-36 weeks of gestation or non-pregnant women will be recruited. As positive controls, healthy pregnant woman at term (over 38 weeks of gestation) will be enrolled. The main outcome assessed is preterm delivery.

ELIGIBILITY:
Inclusion Criteria:

- Singleton pregnancy, monitored in Port Royal or secondarily transferred, between 24 and 32 GA. Hospitalization for preterm labor (cervix < 25 mm at transvaginal cervical ultrasound) or -Singleton pregnancy, monitered in Port Royal between 15-16 weeks of gestation, without complication.

or - Singleton pregnancy, monitered in Port Royal between 35-36 weeks of gestation, without complication.

or - Healthy woman, no pregnancy.

Exclusion Criteria:

* Minor
* Not affiliated to health insurance
* Persons under guardianship or judicial protection
* Infection with HIV, Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV)
* Diabetes or chronic inflammatory disease
* Carrier of B streptococcus
* Cervical strapping
* Fetus with chromosomal abnormalities
* Infections
* Premature rupture of membrane

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2014-12-14 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Delivery | until Day 14
  Assessed among patients in preterm labor between 24 - 32 GA

SECONDARY OUTCOMES:
Delivery before 34 GA | until Day 14
  Assessed among patients in preterm labor between 24 - 32 GA
composite Prenatal maternal care | until Delivery
  Assessed by :
  * number of hospitalization,
  * total duration of hospitalization for preterm labor,
  * use of tocolytic treatment, administration of prenatal corticotherapy,
  * time between the last injection of corticosteroids and birth
composite Neonatal outcome | At Birth
  Assessed by :
  * birth weight,
  * Apgar score at 5 minutes,
  * arterial cord pH,
  * transfer to neonatology unit or neonatal intensive care,
  * death,
  * In case of transfer neonatal unit or neonatal intensive care : duration of hospitalization, use of respiratory assistance
composite Obstetric outcome | At Delivery
  Assessed by :
  * pregnancy term,
  * way to start labor (spontaneous, induction, caesarean before labor)
  * duration of labor,
  * maternal fever,
  * antibiotics during labor,
  * mode of delivery,
  * indications of cesarean

CONTACTS AND LOCATIONS:
Overall Officials: Celine MEHATS, PhD, Study Director — INSERM U1016 - Cochin Hospital Public Hospitals of Paris
Locations (1):
- Maternité Port Royal-Cochin, Paris, France

REFERENCES:
- [Background] Larroque B, Ancel PY, Marret S, Marchand L, Andre M, Arnaud C, Pierrat V, Roze JC, Messer J, Thiriez G, Burguet A, Picaud JC, Breart G, Kaminski M; EPIPAGE Study group. Neurodevelopmental disabilities and special care of 5-year-old children born before 33 weeks of gestation (the EPIPAGE study): a longitudinal cohort study. Lancet. 2008 Mar 8;371(9615):813-20. doi: 10.1016/S0140-6736(08)60380-3. PMID 18328928
- [Background] McLaren J, Malak TM, Bell SC. Structural characteristics of term human fetal membranes prior to labour: identification of an area of altered morphology overlying the cervix. Hum Reprod. 1999 Jan;14(1):237-41. doi: 10.1093/humrep/14.1.237. PMID 10374127
- [Background] Malak TM, Bell SC. Structural characteristics of term human fetal membranes: a novel zone of extreme morphological alteration within the rupture site. Br J Obstet Gynaecol. 1994 May;101(5):375-86. doi: 10.1111/j.1471-0528.1994.tb11908.x. PMID 8018607